CLINICAL TRIAL: NCT06839274
Title: Follicular Volume at the Time of Final Oocyte Maturation in Poor Responders, and Its Correlation With Oocyte Maturity
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2408-ABU-013-AS
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: OVARIAN STIMULATION

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The study population is the infertile patients seeking IVF treatment in ART fertility clinics of Abu: Recruited patients will be stimulated in a antagonist protocol with the use of Pergoveris as gonadotropin with a starting dose of 450 IU. The antagonist will be started on day 5 of the stimulation. Patients will be triggered according to clinical standard protocol for poor ovarian reserve patients when the leading follicle reaches 15 mm (2). The only additional measure will be the measurement of the follicle volumes on the day of trigger and before oocyte pick up procedure. This will be performed at the same time as the pre oocyte pick up ultrasound prior to the patient admission to the recovery room for preparation. The ultrasound that will be used already has a pre build program that calculates the follicular volume automatically and hence not extending the ultrasound time. Oocyte pickup will be performed the same way as per the SOP of the clinic for the patients who have less than 7 follicles on the day of the ovum pickup i.e. each follicle will be punctured, aspirated and then flu
  Interventions: Other: transvaginal Ultrasound

INTERVENTIONS:
Other: transvaginal Ultrasound — The only additional measure will be the measurement of the follicle volumes on the day of trigger and before oocyte pick up procedure. This will be performed at the same time as the pre Oocyte pick up ultrasound prior to the patient admission to the recovery room for preparation. The ultrasound that will be used already has a pre build program that calculates the follicular volume automatically and hence not extending the ultrasound time.

SUMMARY:
Women with a severely diminished ovarian reserve and monofollicular growth are at a higher risk of premature ovulation as well as poor quality oocytes. Our group showed previously that women with severely diminished ovarian reserve benefit from receiving the final oocyte maturation at smaller follicle sizes in terms of reducing the risk of premature ovulation and finding mature oocytes even out of small size follicles.

Adding the measurement of the follicular volume at the time of final oocyte maturation might provide more information on the proper timing of trigger administration compared to the follicular size alone, hormonal profile as well as previous stimulation attempts. Setting a cutoff value of follicular volume for trigger might help to avoid premature ovulation and possibly increase the chances of ending up with a euploid embryo.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age group: 18 -48
* undergoing ovarian stimulation for oocyte vetrification
* undergoing IVF/ ICSI with PGT-A / PGT-M / PGT- Sr
* less than or equal to 3 AFC on initiation of stimulation
* follicular phase stimulation

Exclusion Criteria:

* surgically retrieved sperm

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — * Reproductive age group: 18 -48
  * undergoing ovarian stimulation for oocyte vetrification
  * undergoing IVF/ ICSI with PGT-A / PGT-M / PGT- Sr
  * less than or equal to 3 AFC on initiation of stimulation
  * follicular phase stimulation
Study Population: Patients in ART Fertility Clinics who will undergo ovarian stimulation
  * Reproductive age group: 18 -48
  * undergoing ovarian stimulation for oocyte vetrification
  * undergoing IVF/ ICSI with PGT-A / PGT-M / PGT- Sr
  * less than or equal to 3 AFC on initiation of stimulation
  * follicular phase stimulation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the investigators will see the corellation between the follicular volume at the time of trigger with the oocyte maturity in patients with less than four follicles of a follicle size of at least 11 mm . | 1 year
  The objective of this study is to evaluate the relationship between follicular volume at the time of trigger and oocyte maturity in patients undergoing assisted reproductive techniques, specifically those with fewer than four follicles of at least 11 mm in size. This study aims to determine whether follicular volume just before trigger is a significant predictor of oocyte maturation. By focusing on this specific patient group, the study seeks to provide insights that could inform treatment strategies and improve outcomes in assisted reproductive technology.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Study Director — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
on request